CLINICAL TRIAL: NCT06415279
Title: Clinical Evaluation of the Sebum Reduction Induced by Clascoterone Cream 1%
Brief Title: A Study to Evaluate the Reduction in Sebum (Skin Oil) Induced by Clascoterone Cream 1% in Acne Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCS-67-22
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clascoterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Winlevi (clascoterone) 1% cream (Experimental)
  Interventions: Drug: Winlevi (clascoterone) 1% cream

INTERVENTIONS:
Drug: Winlevi (clascoterone) 1% cream — Twice daily (BID) dosing

SUMMARY:
The etiology of acne is heavily dependent on the production of sebum by the sebaceous glands that results in the growth of the bacteria c. acnes. If no sebum is present, there is no nutritional source for the c. acnes, the bacteria die, and acne resolves. A newly FDA approved acne medication consisting of clascoterone cream 1% is believed to effectively treat acne due to a decrease in sebum production. This mechanism of action has been postulated based on efficacy observed in the phase III trials that lead to its approval. This research aims to demonstrate the effect of clascoterone cream 1% in sebum reduction.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 12+ years of age.
2. Subjects with mild to moderate acne.
3. Subjects must possess 10-100 total non-inflammatory lesions (open comedones and closed comedones), 10-50 total inflammatory lesions, no cysts, and up to 2 nodules (if deemed appropriate by the PI) on the face.
4. Subjects with all Fitzpatrick skin types I-VI.
5. Subjects who agree to use only the study products for acne treatment. No other medicated cleansers or moisturizers or acne treatments of any kind are allowed.
6. Subjects agree not to introduce any new colored cosmetics or skin care products while participating in the study (lipsticks, eye shadows, facial foundations, blush, powder, cleansers, moisturizers).
7. Subjects agree to arrive at all visits with a clean face, having washed his/her face and removed all facial and eye makeup products within 2 hours to 4 hours prior to the visit and is not to use/apply any topical facial product(s) until the visit is completed.
8. No known medical conditions that, in the investigator's opinion, may interfere with study participation.
9. Women of childbearing potential must be willing to use a form of birth control during the study. For the purpose of this study, the following are considered acceptable methods of birth control: oral contraceptives, Norplant, Depo-Provera, double barrier methods (e.g., condom and spermicide) and abstinence.
10. Subjects are dependable and able to follow directions and willing to comply with the schedule of visits.
11. Subjects in generally good physical and mental health.
12. Able to read, write, speak, and understand English
13. Individual (and/or his/her legally acceptable representative, as applicable) has signed the Consent for Photograph Release and ICD (and/or Assent Document, as applicable) including Health Insurance Portability and Accountability Act (HIPAA) disclosure.
14. Subject must avoid sun exposure, or use sunscreen if sun exposure is unavoidable.
15. Subject must avoid professional or facial spa procedures during the study.

Exclusion Criteria:

1. Any dermatological disorder, which in the investigator's opinion, may interfere with the accurate evaluation of the subject's skin characteristics, except for the study condition of acne.
2. Subjects who are not willing to use the assigned study product to their face as instructed.
3. Subjects who have acne nodules/cysts representative of severe acne.
4. Subjects who are currently using, planning to use during the study or has used any of the following in the specified time range (based on subject report):

   * 1 month prior to Visit 1: Prescription (oral or topically applied on the face) antibiotics, inhaled steroids (except those prescribed for allergies), or hormones (pre- or post-menopausal hormone-replacement therapy; insulin, etc.), or other medications that could make skin more sensitive or have an effect on the skin, as determined by the PI or designee. Oral contraceptives are acceptable.
   * 1 month prior to Visit 1: Prescription medication for acne (e.g. doxycycline, minocycline, clindamycin, sulfamethoxazole and trimethoprim [Bactrim], tetracycline, erythromycin, azithromycin, or Vibramycin®)
   * 1 month prior to Visit 1: Topical prescription retinoids (e.g. Retin-A®, Retin-A Micro®, Renova®, Adapalene, Tazarotene, Avita®, Tazorac®, Avage®, Differin®), azelaic acid, benzoyl peroxide, dapsone, sodium sulfacetamide, Epiduo®, or other similar prescription drug on the face
   * 6 months prior to Visit 1: Accutane or other oral retinoid
   * 2 weeks prior to Visit 1: Any of the following on the face:

     * Light therapy
     * OTC topical medications/products (including antiacne or antibacterial agents, topical anti-inflammatories, topical retinoids, etc.). Sunscreens (SPF) are acceptable.
5. Females who are pregnant, lactating, or planning to become pregnant during the study or within 30 days of study completion. (Subject must document her response in either the source documentation or informed consent/assent forms).
6. Subject has a surgery and/or invasive medical procedure planned during the study.
7. Subject has observable suntan, scars, nevi, tattoo, excessive hair (including beard, mustache, or goatee), or other dermal conditions on the face that that could interfere with study evaluations or confound study results, as determined by the PI or designee.
8. Subject is taking medications that would mask an adverse event (AE) or influence the study results, including:

   * Immunosuppressive drugs and steroidal and/or non-steroidal anti-inflammatory drugs within 3 months before Visit 1 and during the study.
   * Regular use of antihistamines within 1 month before Visit 1 and during the study.
9. Subject has a history of or a concurrent health condition/situation, which in the opinion of the PI, if medically qualified, or Study Physician, may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study.
10. Subject is an employee/contractor or immediate family member of the PI, Study Site, or Sponsor.
11. Subjects with clinically significant unstable medical disorders.
12. Subjects who are unwilling or unable to comply with the requirements of the protocol.
13. Subjects with any known allergies or sensitivities to the study acne products.
14. Subjects who are currently under the care of a dermatologist for acne.
15. Subjects who are currently experiencing an acne flare.
16. Subjects who have history of a psychological illness or condition that would interfere with their ability to understand and follow the requirements of the study.
17. Subjects having started hormone replacement therapies (HRT) or hormones for birth control less than 3 months prior to the study entry or who plan on starting, stopping or changing doses of HRT or hormones for birth control during the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the change in causal sebum measurements from the forehead obtained with a sebumeter during the study. | Weeks 16

SECONDARY OUTCOMES:
The secondary efficacy endpoint is the changes in the facial microbiome induced by 8, 12, and 52 weeks of clascoterone 1% cream application. | Weeks 52

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Consulting Services, PLLC, High Point, North Carolina, United States

REFERENCES:
- [Derived] Draelos ZD, Kyeremateng K, Squittieri N. Reduction in Facial Sebum Production Following Treatment with Clascoterone Cream 1% in Patients with Acne Vulgaris: 12-Week Interim Analysis. Dermatol Ther (Heidelb). 2025 Sep;15(9):2657-2666. doi: 10.1007/s13555-025-01495-y. Epub 2025 Jul 19. PMID 40682762